CLINICAL TRIAL: NCT02575092
Title: Department of Geriatrics
Brief Title: The Relationship Between HHcy and Contrast-induced Nephropathy in Hypertensive Patients After Coronary Artery Diagnosis and Treatment
Acronym: CONTRAST-CADT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fuling Central Hospital of Chongqing City (Other)
Responsible Party: Principal Investigator, Lu Jian-gang,MD, Department of Geriatrics, Fuling Central Hospital of Chongqing City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lu 20143440
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Homocysteine; Coronary Disease; Angioplasty,Balloon,Coronary; Contrast Media; Nephropathy; Hypertension
Keywords: Hyperhomocysteinemia; Coronary angiography; Percutaneous coronary intervention; Hypertension; Contrast-induced nephropathy
MeSH Terms: conditions — Coronary Disease; Kidney Diseases; Hypertension; Hyperhomocysteinemia | interventions — Enalapril

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A, without hypertension (Active Comparator): The patients who will not be taken the drugs of antihypertension and antihomocysteine.
  Interventions: Drug: Placebo
- Group B, hypertension (Experimental): The hypertensive patients with their plasma Hcy levels <10 umol/L will be taken the drugs of antihypertension(Enalapril Maleate Tablets,as the program-based antihypertension)
  Interventions: Drug: Enalapril Maleate Tablets(as the program-based antihypertension)
- Group C,hypertension and hyperhomocysteinemia (Experimental): The hypertensive patients with their plasma Hcy levels ≥10 umol/L will be taken the drugs of antihypertension and antihomocysteine( Enalapril Maleate and Folic Acid Tablets,as the program-based antihypertension)
  Interventions: Drug: Enalapril Maleate and Folic Acid tablets(as the program-based antihypertension)

INTERVENTIONS:
Drug: Enalapril Maleate Tablets(as the program-based antihypertension)
  Arms: Group B, hypertension
Drug: Enalapril Maleate and Folic Acid tablets(as the program-based antihypertension)
  Arms: Group C,hypertension and hyperhomocysteinemia
Drug: Placebo
  Arms: Group A, without hypertension

SUMMARY:
Contrast-induced nephropathy has become the third-largest cause of hospital acquired acute renal injury, and which morbidity is only less than that of renal hypoperfusion and renal toxicity of drugs, about 11%of all cases. Pathophysiologic mechanisms of contrast-induced nephropathy(CIN) is not entirely clear yet. May be associated with renal hemodynamic changes, medullary ischemia because of renal blood flow reduction, oxidative stress, endothelial dysfunction ,contrast agents damage the epithelium of renal tubular directly and so on. Currently the studies have proved that inflammation(CRP, TNF-α and NF-қB) played a role in CIN.It is well-know that the hyperhomocysteinemia(HHCY) is a independent risk factor for cardiovascular diseases, which has pro-inflammatory effects. Researches showed that Hcy stimulated CRP generation by the NMDAr-ROS-ERK1 / 2 / p38-NF-қB signaling pathway and triggered inflammatory response. We will compare the CIN incidence of different plasma Hcy levels in adults hypertensive patients undergoing coronary artery diagnosis and treatment(CAG and PCI). CIN was defined as an absolute ≥0.5mg/dl or a relative ≥25% increase in the serum creatinine level at 48 hours after the procedure. The relationship between decreased plasma Hcy levels and blood pressure values by using Enalapril Maleate and Folic Acid Tablets(as the program-based antihypertension) and recovery of CIN has been observed. Using univariate and multivariate Logistic regression to analyse the relationship between HHcy and CIN, and taking receiver operating characteristic (ROC) curve to select the best Hcy plasma levels that which can predict the CIN and the probability. This study will help us to understand the relationship between HHcy and CIN that course of the procedure in adults hypertensive patients, preoperative plasma Hcy levels can predict the incidence of CIN and whether Enalapril Maleate Folic Acid tablets can reduce the CIN of hypertensive patients with HHcy. Which has important clinical significance. This study also offer feasibility for further research that HHcy plays a role in pathogenesis and specific signaling pathways of CIN.

DETAILED DESCRIPTION:
The first stage: the establishment of hypothesis of the relationship between HHcy and CIN The demographic and laboratory data were retrieved from the His system. Hypertensive patients who underwent coronary artery diagnosis and treatment(CAG or PCI) at Fuling Central Hospital of Chongqing City from June 2013 to August 2015 were initially included in the present study. The baseline characteristics of the hypertensive patients according to the tertile of plasma homocysteine level will be analysed, and investigating the incidence of CIN and relevant factors.

The second stage: To verify the hypothesis of relationship between HHcy and CIN in patients with hypertension CER research method

1. patients who accepted the coronary artery diagnosis and treatment(CAG and PCI ) in departments of Geriatrics and Cardiovascular within one year were initially participate in. According to the statistics that we finished, the proportion of hypertension in the total patients who underwent procedure has reached about 80%, so there has more than 4000 patients with hypertension within 1 year will be involved. The levels of plasma Hcy in the total patients will be detected. The patients will divided into 2 groups according to the plasma Hcy levels,The hypertensive patients(adults) with their plasma Hcy levels ≥10 umol/L will take Enalapril Maleate and Folic Acid Tablets(as the program-based antihypertension), The hypertensive patients(adults) with their plasma Hcy levels <10 umol/L will take Enalapril Maleate Tablets(as the program-based antihypertension).The procedure will be carried out after blood pressure valves within normal range.
2. All patients will be followed up for 3 months, they will return to hospital 3 times(once a month) after discharged. Urine routine and renal function will be tested, to register blood pressure,any change of body condition and other related factors per months, and plasma Hcy levels will be detected in the hypertensive patients with higher-homocysteinemia at second and third months after discharged.
3. Data collection and data statistics will be carried out per 2 months. All patients who undergoing coronary artery diagnosis and treatment(CAG and PCI)will be divided into group A without hypertension, group B that the hypertensive patients with their plasma Hcy levels <10 umol/L and group C that the hypertensive patients with plasma Hcy levels ≥10 umol/L. To compare CIN incidence of the 3 groups at each time point, the CIN incidence of group B and group C will be compared, and association between CIN and the levels of blood pressure and plasma Hcy will be analyzed by multivariate logistic regression analysis according to the ROC curve.

ELIGIBILITY:
Inclusion Criteria:

From November 2015 to April 2017 , all consecutive patients admitted to the participating centers for the patients who undergoing coronary artery diagnosis and treatment(CAG or PCI) will been considered eligible，about 5500 cases.

Exclusion Criteria:

* Who requires long-term peritoneal or hemodialysis.
* Who had been underwent a kidney transplantation.
* Renal failure with a creatinine level >3 mg/dl.
* Who had been received the contrast agent within 2 weeks or had been received metformin, aminoglycoside antibiotics or acetylcysteine within 48 hours.
* Iodine allergy, acute and chronic infections and hyperthyroidism.
* Left ventricular ejection fraction <30%.
* Secondary hypertension.
* Who can not be tolerated ACEI.
* Any other surgical contraindications.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The incidence of contrast-induced nephropathy | At 48 hours after the procedure.
  CIN was defined as an absolute ≥0.5mg/dl or a relative ≥25% increase in the serum creatinine level at 48 hours after the procedure.

SECONDARY OUTCOMES:
Dialysis | Within the first 3 months after procedure.
  The hypertensive patients in the 3 groups who had been diagnosed as CIN need to dialysis.
Ischemic stroke | Within the first 3 months after procedure.
  The hypertensive patients in the 3 groups who had been diagnosed of ischemic stroke (focal neurological deficits persisting for more than 24 hours) confirmed by non-investigational CT or MRI
All cause mortality | Within the first 3 months after procedure.
  Any cause of death in patients

CONTACTS AND LOCATIONS:
Locations (1):
- TIAN Jie, Fuling, Chongqing Municipality, China

REFERENCES:
- [Result] Kim SJ, Choi D, Ko YG, Kim JS, Han SH, Kim BK, Kang SW, Hong MK, Jang Y, Choi KH, Yoo TH. Relation of homocysteinemia to contrast-induced nephropathy in patients undergoing percutaneous coronary intervention. Am J Cardiol. 2011 Oct 15;108(8):1086-91. doi: 10.1016/j.amjcard.2011.06.010. Epub 2011 Jul 24. PMID 21791335
- [Result] Bolognese L, Falsini G, Grotti S, Limbruno U, Liistro F, Carrera A, Angioli P, Picchi A, Ducci K, Pierli C. The contrast media and nephrotoxicity following coronary revascularization by primary angioplasty for acute myocardial infarction study: design and rationale of the CONTRAST-AMI study. J Cardiovasc Med (Hagerstown). 2010 Mar;11(3):199-206. doi: 10.2459/JCM.0b013e32833186a4. PMID 19829124